CLINICAL TRIAL: NCT00575159
Title: A Double-blind, Randomized, Single Ascending Dose Escalation, Placebo-controlled, Crossover Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK189075 Administered to Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Assess the Safety of Single Doses of GSK189075 in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KGI107465
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 Diabetes mellitus, pharmacokinetics,; pharmacodynamics; Adult male and females,
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm a (Experimental): GSK189075
  Interventions: Drug: GSK189075
- Arm b (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GSK189075 — investigational drug
  Arms: Arm a
Drug: placebo — placebo comparator
  Other Names: GSK189075
  Arms: Arm b

SUMMARY:
The purpose of this research study is to look at concentrations of GSK189075 in blood when single doses of the drug are taken by mouth in combination with basal insulin. The clinical effects of the drug in combination with insulin on the body will also be studied. The results will help determine doses of GSK189075 can be studied in the future in the type I diabetes mellitus population.

ELIGIBILITY:
Inclusion Criteria:

* Adult male/female, 18 to 55 years old
* Diagnosis of type 1 diabetes mellitus for at least 6 months; and using a continuous insulin pump
* Willing and able to follow all study-related instructions provided by the site staff.
* Willing to provide signed informed consent.

Exclusion Criteria:

* Pregnant or a nursing female.
* Have a past or current disease such as heart, liver, kidney, blood, brain, or other disease.
* Have HIV or hepatitis, or have alcohol or drugs in your system at the screening visit.
* Have a history of alcohol abuse or have an eating disorder
* Have been in another research study in the last month or have taken certain medications in the 1 week before study drug would be taken.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2008-12-18 (Actual); Study Completion 2008-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, San Diego, California, United States

REFERENCES:
- [Derived] Mudaliar S, Armstrong DA, Mavian AA, O'Connor-Semmes R, Mydlow PK, Ye J, Hussey EK, Nunez DJ, Henry RR, Dobbins RL. Remogliflozin etabonate, a selective inhibitor of the sodium-glucose transporter 2, improves serum glucose profiles in type 1 diabetes. Diabetes Care. 2012 Nov;35(11):2198-200. doi: 10.2337/dc12-0508. Epub 2012 Sep 25. PMID 23011728

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 participants with type 1 diabetes mellitus (T1DM) were randomized in this study. Study was conducted between 31 Mach 2008 to 19 January 2009 at a single center in the United States (US).
Pre-assignment Details: Participants were screened within 28 days of the first dose and a total of 10 participants were randomized to receive the study drug. The participants were admitted on Day -2 and were analyzed of all Baseline safety and glucose control on Day -1.
Groups:
- Overall Study Arm: Participants received 5 treatments P0, P1, A, B, C in each of the treatment period in a randomized manner separated by a 5 to 35-day washout period between treatments, where Treatment P0 consisted of Basal insulin [continuous subcutaneous insulin injection (CSII)], mealtime placebo injection, and placebo tablet. Treatment P1 consisted of CSII, mealtime bolus insulin injection, and Placebo tablet. Treatment A consisted of CSII, mealtime placebo injection, GSK189075 50 milligram (mg) tablet. Treatment B consisted of CSII, mealtime placebo injection, GSK189075 150 mg tablet. Treatment C consisted of CSII, mealtime placebo injection, GSK189075 500 mg tablet. The two placebo sessions (P0 and P1) were designed to provide information about the relative efficacy of GSK189075 versus each individual participant's usual mealtime insulin bolus. The number of tablets administered will be same for each treatment arm.
Period: Overall Study
Arm/Group | Overall Study Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Arm: Participants received 5 treatments P0, P1, A, B, C in each of the treatment period in a randomized manner separated by a 5 to 35-day washout period between treatments, where Treatment P0 consisted of Basal insulin [continuous subcutaneous insulin injection (CSII)], mealtime placebo injection, and placebo tablet. Treatment P1 consisted of CSII, mealtime bolus insulin injection, and Placebo tablet. Treatment A consisted of CSII, mealtime placebo injection, GSK189075 50 mg tablet. Treatment B consisted of CSII, mealtime placebo injection, GSK189075 150 mg tablet. Treatment C consisted of CSII, mealtime placebo injection, GSK189075 500 mg tablet. The two placebo sessions (P0 and P1) were designed to provide information about the relative efficacy of GSK189075 versus each individual participant's usual mealtime insulin bolus. The number of tablets administered will be same for each treatment arm.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to 6 months
Population: Safety Population comprised of all enrolled participants who have received at least one dose of study drug were included in the safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received a single dose of Basal insulin (CSII), mealtime placebo injection and matching GSK189075 placebo tablet. On Day 1, all study doses and mealtime insulin boluses were administered 15 minutes before the Participant begins to eat the scheduled meal (on dosing day, breakfast was the oral glucose load; lunch was the standard meal). On Day -1 (day prior to dosing day), basal insulin and insulin boluses before each meal were administered by the continuous insulin infusion pump. Study medication was administered orally in a fasted state before breakfast with 250 milliliter (mL) of water.
- Placebo+ Prandial Insulin: Participants received a single dose of Basal insulin (CSII), mealtime bolus insulin injection and matching GSK189075 placebo tablet. On Day 1, all study doses and mealtime insulin boluses were administered 15 minutes before the Participant begins to eat the scheduled meal (on dosing day, breakfast was the oral glucose load; lunch was the standard meal). On Day -1 (day prior to dosing day), basal insulin and insulin boluses before each meal were administered by the continuous insulin infusion pump. Study medication was administered orally in a fasted state before breakfast with 250mL of water.
- GSK189075 50mg: Participants received a single dose of Basal insulin (CSII), mealtime placebo injection and GSK189075 50 mg tablet. On Day 1, all study doses and mealtime insulin boluses were administered 15 minutes before the Participant begins to eat the scheduled meal (on dosing day, breakfast was the oral glucose load; lunch was the standard meal). On Day -1 (day prior to dosing day), basal insulin and insulin boluses before each meal were administered by the continuous insulin infusion pump. Study medication was administered orally in a fasted state before breakfast with 250mL of water.
- GSK189075 150mg: Participants received a single dose of Basal insulin (CSII), mealtime placebo injection and GSK189075 150 mg tablet. On Day 1, all study doses and mealtime insulin boluses were administered 15 minutes before the Participant begins to eat the scheduled meal (on dosing day, breakfast was the oral glucose load; lunch was the standard meal). On Day -1 (day prior to dosing day), basal insulin and insulin boluses before each meal were administered by the continuous insulin infusion pump. Study medication was administered orally in a fasted state before breakfast with 250mL of water.
- GSK189075 500mg: Participants received a single dose of Basal insulin (CSII), mealtime placebo injection and GSK189075 500 mg tablet. On Day 1, all study doses and mealtime insulin boluses were administered 15 minutes before the Participant begins to eat the scheduled meal (on dosing day, breakfast was the oral glucose load; lunch was the standard meal). On Day -1 (day prior to dosing day), basal insulin and insulin boluses before each meal were administered by the continuous insulin infusion pump. Study medication was administered orally in a fasted state before breakfast with 250mL of water.
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Any AE | 3 | 4 | 5 | 6 | 4
  Any SAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Hypoglycemia Episodes/Events
Description: A hypoglycemic event was defined as symptoms of hypoglycemia confirmed by a blood glucose value below normal limits [less than 3.89 millimoles per liter (mmol/L)] or 70 milligrams per deciliter (mg/dL). Symptoms of hypoglycemia without confirmed blood glucose values were reported as AEs instead of hypoglycemic events. Number of participants with hypoglycemic events were reported.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received a single dose of Basal insulin (CSII), mealtime placebo injection and matching GSK189075 placebo tablet. On Day 1, all study doses and mealtime insulin boluses were administered 15 minutes before the Participant begins to eat the scheduled meal (on dosing day, breakfast was the oral glucose load; lunch was the standard meal). On Day -1 (day prior to dosing day), basal insulin and insulin boluses before each meal were administered by the continuous insulin infusion pump. Study medication was administered orally in a fasted state before breakfast with 250mL of water.
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 5 | 5 | 3 | 5 | 6

3. Primary Outcome: Change From Baseline Vital Signs: Systolic and Diastolic Blood Pressure (SBP and DBP)
Description: SBP and DBP were obtained during each treatment period at the indicated time points. Measurements were made with the participant lying semi-recumbent having rested in this position for at least 10 minute before the initial reading.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Millimeters of mercury (mmHg)
  SBP,Day1,0.5 H | 1.6 (10.63) | -5.1 (5.32) | -0.7 (18.03) | -3.4 (12.97) | -1.9 (8.82)
  SBP,Day1,1 H | 1.8 (14.70) | -1.7 (9.17) | -4.7 (12.78) | -7.8 (8.77) | 5.6 (14.75)
  SBP,Day1,2 H | -1.8 (14.01) | -6.5 (6.29) | -5.1 (14.30) | -3.5 (13.19) | -2.2 (9.38)
  SBP,Day1,4 H | -2.9 (11.86) | -0.9 (7.56) | -8.4 (8.37) | -2.5 (18.52) | -4.3 (7.49)
  SBP,Day1,6 H | -2.1 (9.88) | -5.5 (13.10) | -8.2 (7.18) | -8.4 (15.43) | -6.9 (13.58)
  SBP,Day1,8 H | -1.4 (13.12) | -2.1 (10.80) | -3.2 (10.21) | -7.3 (18.50) | -2.4 (12.56)
  SBP,Day1,24 H | 2.6 (7.27) | -1.4 (11.77) | -0.4 (9.54) | -0.2 (12.20) | -4.6 (12.85)
  DBP,Day1,0.5 H | -1.1 (10.36) | -5.3 (9.38) | -9.8 (11.73) | -7.4 (13.13) | -5.2 (13.36)
  DBP,Day1,1 H | -5.4 (11.61) | -7.7 (12.31) | -11.5 (8.32) | -15.1 (11.06) | -5.7 (9.59)
  DBP,Day1,2 H | -8.8 (7.50) | -8.7 (11.29) | -11.7 (10.04) | -11.0 (12.72) | -7.2 (10.55)
  DBP,Day1,4 H | -6.4 (7.52) | -6.4 (13.08) | -11.7 (7.45) | -8.5 (13.04) | -7.7 (9.84)
  DBP,Day1,6 H | -8.4 (8.88) | -7.0 (10.70) | -13.2 (8.31) | -12.3 (15.36) | -8.0 (12.91)
  DBP,Day1,8 H | -2.2 (7.79) | -5.8 (9.24) | -10.1 (5.76) | -10.7 (15.40) | -4.7 (15.05)
  DBP,Day1,24 H | 0.5 (9.97) | 1.6 (11.55) | -4.2 (6.71) | -3.6 (11.51) | -2.0 (9.51)

4. Primary Outcome: Change From Baseline Vital Signs: Heart Rate
Description: Heart rate was obtained during each treatment period at indicated time points. Measurements were made with the participants lying semi-recumbent having rested in this position for at least 10 minutes before the initial reading.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
beats/minute
  Day 1,0.5 H | -1.4 (9.69) | -5.4 (8.57) | -4.5 (7.21) | -4.7 (7.58) | -5.2 (12.67)
  Day 1,1 H | 1.7 (11.46) | -2.8 (8.65) | -1.4 (8.23) | -4.3 (11.20) | -5.1 (12.96)
  Day 1,2 H | 1.0 (13.79) | -4.0 (7.90) | -4.4 (8.22) | -3.3 (7.42) | -5.1 (14.05)
  Day 1,4 H | -1.4 (11.37) | -4.6 (10.46) | -6.5 (7.94) | -2.6 (9.79) | -6.8 (10.90)
  Day 1,6 H | 2.5 (11.20) | -2.0 (8.46) | -1.3 (10.36) | 3.5 (11.54) | -1.4 (12.17)
  Day 1,8 H | 0.7 (12.48) | -6.6 (10.60) | -4.6 (6.95) | 1.6 (10.16) | -3.4 (12.04)
  Day 1,24 H | 5.4 (13.92) | 6.6 (11.67) | 4.2 (10.99) | 10.0 (11.50) | 0.4 (12.39)

5. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Standard semi-recumbent 12-lead ECG was obtained after the participant rested for a minimum of 10 minutes (If questionable abnormality was noted on the ECG, 2 more measurements were allowed to provide an average of 3 measurements). Number of participants with abnormal ECG were reported.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  DAY -2 | 0 | 1 | 1 | 3 | 0
  DAY -2 (2) | 0 | 0 | 1 | 2 | 0
  DAY -2 (3) | 0 | 1 | 1 | 2 | 0
  DAY -1 | 1 | 0 | 0 | 0 | 0
  DAY -1 (2) | 1 | 0 | 1 | 0 | 0
  DAY -1 (3) | 1 | 0 | 0 | 0 | 0
  DAY 1 PRE-DOSE | 1 | 3 | 3 | 2 | 3
  DAY 1 PRE-DOSE (2) | 1 | 3 | 3 | 3 | 3
  DAY 1 PRE-DOSE (3) | 1 | 3 | 3 | 3 | 3
  DAY 1 4 H | 2 | 1 | 2 | 3 | 3
  DAY 1 24 H | 2 | 0 | 1 | 2 | 1

6. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Data
Description: Clinical Chemistry data for parameters: Alanine Amino Transferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Bicarbonate, Calcium, Chloride, Creatine Kinase, Creatinine, Gamma Glutamyl Transferase (GGT), Glucose, Lactate Dehydrogenase, Magnesium, Phosphorus, Potassium, Total Bilirubin, Sodium, Total protein, triglycerides and urea/BUN was reported. Data for number of participants with abnormal clinical Chemistry data was presented.
Time Frame: Day 1 of each treatment period
Population: Safety Population. Only those participants available at the specific time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  ALT,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 5 | 6 | 7 | 6 | 6
  ALT,DAY 1, PRE-DOSE,Normal | 4 | 5 | 6 | 6 | 5
  ALT,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 2 | 6 | 7 | 6 | 6
  ALT,DAY 1 ,PRE-DOSE,Low | 1 | 1 | 1 | 0 | 1
  ALT,DAY 1, 24 H,Normal: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  ALT,DAY 1, 24 H,Normal | 8 | 8 | 7 | 6 | 7
  ALT,DAY 1, 24 H,Low: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  ALT,DAY 1, 24 H,Low | 2 | 1 | 2 | 1 | 2
  ALT,DAY 1, 24 H,Missing: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  ALT,DAY 1, 24 H,Missing | 0 | 1 | 1 | 1 | 1
  Albumin,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Albumin,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Albumin,DAY 1, 24 H,High | 1 | 0 | 1 | 0 | 0
  Albumin,DAY 1, 24 H,Normal | 9 | 10 | 9 | 10 | 10
  ALP,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  ALP,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  ALP,DAY 1, 24 H,Normal | 10 | 10 | 10 | 10 | 10
  AST,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 5 | 6 | 7 | 6 | 6
  AST,DAY 1, PRE-DOSE,Normal | 5 | 6 | 6 | 5 | 6
  AST,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 5 | 6 | 7 | 6 | 6
  AST,DAY 1 ,PRE-DOSE,Low | 0 | 0 | 1 | 1 | 0
  AST,DAY 1, 24 H,Normal: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  AST,DAY 1, 24 H,Normal | 9 | 9 | 6 | 6 | 8
  AST,DAY 1, 24 H,Low: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  AST,DAY 1, 24 H,Low | 1 | 1 | 3 | 2 | 2
  AST,DAY 1, 24 H,Missing: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  AST,DAY 1, 24 H,Missing | 0 | 0 | 1 | 0 | 0
  Bicarbonate,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Bicarbonate,DAY 1, PRE-DOSE,Normal | 6 | 6 | 6 | 6 | 6
  Bicarbonate,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Bicarbonate,DAY 1 ,PRE-DOSE,Low | 0 | 0 | 1 | 0 | 0
  Calcium,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Calcium,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Chloride,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Chloride,DAY 1, PRE-DOSE,High | 1 | 0 | 0 | 0 | 0
  Chloride,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Chloride,DAY 1, PRE-DOSE,Normal | 5 | 6 | 7 | 6 | 6
  Chloride,DAY 1, 24 H,Normal | 10 | 10 | 10 | 10 | 10
  Creatine Kinase,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Creatine Kinase,DAY 1, PRE-DOSE,High | 2 | 2 | 2 | 1 | 1
  Creatine Kinase,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Creatine Kinase,DAY 1, PRE-DOSE,Normal | 4 | 4 | 5 | 5 | 5
  Creatinine,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Creatinine,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Creatinine,DAY 1, 24 H,Normal | 10 | 10 | 10 | 10 | 10
  GGT,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6
  GGT,DAY 1, PRE-DOSE,Normal | 5 | 5 | 5 | 6 | 6
  GGT,DAY 1, PRE-DOSE,Missing: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6
  GGT,DAY 1, PRE-DOSE,Missing | 0 | 0 | 1 | 0 | 0
  GGT,DAY 1, 24 H,Normal: number analyzed (Participants) | 10 | 10 | 9 | 10 | 10
  GGT,DAY 1, 24 H,Normal | 10 | 10 | 9 | 10 | 10
  Glucose,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Glucose,DAY 1, PRE-DOSE,High | 3 | 5 | 4 | 3 | 0
  Glucose,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Glucose,DAY 1, PRE-DOSE,Normal | 2 | 1 | 3 | 3 | 6
  Glucose,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Glucose,DAY 1 ,PRE-DOSE,Low | 1 | 0 | 0 | 0 | 0
  Glucose,DAY 1, 24 H,High | 7 | 8 | 6 | 7 | 7
  Glucose,DAY 1, 24 H,Normal | 3 | 2 | 3 | 3 | 3
  Glucose,DAY 1, 24 H,Low | 0 | 0 | 1 | 0 | 0
  Lactate Dehydrogenase,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 5 | 5 | 6 | 4 | 5
  Lactate Dehydrogenase,DAY 1, PRE-DOSE,Normal | 5 | 5 | 6 | 4 | 5
  Magnesium,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Magnesium,DAY 1, PRE-DOSE,Normal | 6 | 6 | 6 | 6 | 6
  Phosphorus, inorganic,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Phosphorus, inorganic,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Potassium,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Potassium,DAY 1, PRE-DOSE,High | 0 | 0 | 1 | 0 | 0
  Potassium,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Potassium,DAY 1, PRE-DOSE,Normal | 6 | 6 | 6 | 6 | 6
  Potassium,DAY 1, 24 H,Normal: number analyzed (Participants) | 10 | 10 | 10 | 8 | 10
  Potassium,DAY 1, 24 H,Normal | 10 | 10 | 10 | 8 | 10
  Sodium,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Sodium,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Sodium,DAY 1, 24 H,Normal | 10 | 10 | 10 | 10 | 10
  Total Bilirubin,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Bilirubin,DAY 1, PRE-DOSE,Normal | 6 | 6 | 6 | 5 | 6
  Total Bilirubin,DAY 1, PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Bilirubin,DAY 1, PRE-DOSE,Low | 0 | 0 | 1 | 1 | 0
  Total Bilirubin,DAY 1, 24 H,Normal | 10 | 10 | 10 | 10 | 10
  Total Protein,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Protein,DAY 1, PRE-DOSE,Normal | 4 | 5 | 5 | 4 | 5
  Total Protein,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Protein,DAY 1 ,PRE-DOSE,Low | 2 | 1 | 2 | 2 | 1
  Total Protein,DAY 1, 24 H,Normal | 9 | 9 | 10 | 9 | 10
  Total Protein,DAY 1, 24 H,Low | 1 | 1 | 0 | 1 | 0
  Triglycerides,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Triglycerides,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Urea/BUN,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Urea/BUN,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Urea/BUN,DAY 1, 24 H,Normal | 10 | 8 | 10 | 10 | 10
  Urea/BUN,DAY 1, 24 H,Low | 0 | 2 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Hematology Data
Description: Data for abnormal Hematology parameters: Basophils, Eosinophils, Hematocrit, Hemoglobin, Lymphocytes, Mean Corpuscle Hemoglobin (MCH), Mean Corpuscle Volume (MCV), Monocytes, Platelet count, Red Blood Cell (RBC), Reticulocytes, Total Neutrophils, White Blood Cell (WBC) were reported. Data for number of participants with abnormal Hematology were reported.
Time Frame: Day 1 of each treatment period
Population: Safety Population. Only those participants available at the specific time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Basophils,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 5 | 7 | 6 | 6
  Basophils,DAY 1, PRE-DOSE,High | 1 | 0 | 2 | 1 | 0
  Basophils,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 5 | 7 | 6 | 6
  Basophils,DAY 1, PRE-DOSE,Normal | 5 | 5 | 5 | 5 | 6
  Basophils,DAY 1, 24 H,High: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Basophils,DAY 1, 24 H,High | 2 | 1 | 0 | 0 | 2
  Basophils,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Basophils,DAY 1, 24 H,Normal | 7 | 8 | 9 | 9 | 8
  Eosinophils,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Eosinophils,DAY 1, PRE-DOSE,High | 5 | 5 | 5 | 5 | 6
  Eosinophils,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Eosinophils,DAY 1, PRE-DOSE,Normal | 1 | 1 | 2 | 1 | 0
  Eosinophils,DAY 1, 24 H,High: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Eosinophils,DAY 1, 24 H,High | 5 | 4 | 4 | 4 | 7
  Eosinophils,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Eosinophils,DAY 1, 24 H,Normal | 4 | 5 | 5 | 5 | 3
  Hematocrit,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Hematocrit,DAY 1, PRE-DOSE,Normal | 2 | 1 | 4 | 2 | 2
  Hematocrit,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Hematocrit,DAY 1 ,PRE-DOSE,Low | 4 | 5 | 3 | 4 | 4
  Hematocrit,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  Hematocrit,DAY 1, 24 H,Normal | 4 | 6 | 7 | 8 | 6
  Hematocrit,DAY 1, 24 H,Low: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  Hematocrit,DAY 1, 24 H,Low | 5 | 4 | 2 | 1 | 4
  Hemoglobin,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Hemoglobin,DAY 1, PRE-DOSE,Normal | 4 | 4 | 6 | 5 | 5
  Hemoglobin,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Hemoglobin,DAY 1 ,PRE-DOSE,Low | 2 | 2 | 1 | 1 | 1
  Hemoglobin,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  Hemoglobin,DAY 1, 24 H,Normal | 7 | 8 | 7 | 8 | 8
  Hemoglobin,DAY 1, 24 H,Low: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  Hemoglobin,DAY 1, 24 H,Low | 2 | 2 | 2 | 1 | 2
  Lymphocytes,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Lymphocytes,DAY 1, PRE-DOSE,Normal | 6 | 6 | 6 | 6 | 6
  Lymphocytes,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Lymphocytes,DAY 1 ,PRE-DOSE,Low | 0 | 0 | 1 | 0 | 0
  Lymphocytes,DAY 1, 24 H,High: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Lymphocytes,DAY 1, 24 H,High | 0 | 0 | 1 | 0 | 0
  Lymphocytes,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Lymphocytes,DAY 1, 24 H,Normal | 9 | 8 | 8 | 7 | 9
  Lymphocytes,DAY 1, 24 H,Low: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Lymphocytes,DAY 1, 24 H,Low | 0 | 1 | 0 | 2 | 1
  MCH,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  MCH,DAY 1, PRE-DOSE,High | 4 | 3 | 4 | 2 | 2
  MCH,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  MCH,DAY 1, PRE-DOSE,Normal | 2 | 3 | 3 | 4 | 4
  MCHC,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  MCHC,DAY 1, PRE-DOSE,High | 4 | 4 | 5 | 5 | 3
  MCHC,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  MCHC,DAY 1, PRE-DOSE,Normal | 2 | 2 | 2 | 1 | 3
  MCV,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  MCV,DAY 1, PRE-DOSE,High | 1 | 1 | 2 | 1 | 1
  MCV,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  MCV,DAY 1, PRE-DOSE,Normal | 5 | 5 | 5 | 5 | 5
  Monocytes,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Monocytes,DAY 1, PRE-DOSE,High | 2 | 2 | 2 | 3 | 2
  Monocytes,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Monocytes,DAY 1, PRE-DOSE,Normal | 4 | 4 | 5 | 3 | 4
  Monocytes,DAY 1, 24 H,High: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Monocytes,DAY 1, 24 H,High | 0 | 1 | 1 | 1 | 1
  Monocytes,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Monocytes,DAY 1, 24 H,Normal | 9 | 8 | 8 | 8 | 9
  Platelet count,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Platelet count,DAY 1, PRE-DOSE,Normal | 6 | 6 | 7 | 6 | 6
  Platelet count,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  Platelet count,DAY 1, 24 H,Normal | 9 | 10 | 9 | 8 | 10
  Platelet count,DAY 1, 24 H,Low: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  Platelet count,DAY 1, 24 H,Low | 0 | 0 | 0 | 1 | 0
  RBC,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  RBC,DAY 1 ,PRE-DOSE,Low | 6 | 6 | 7 | 6 | 6
  RBC,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  RBC,DAY 1, 24 H,Normal | 2 | 2 | 3 | 4 | 1
  RBC,DAY 1, 24 H,Low: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  RBC,DAY 1, 24 H,Low | 7 | 8 | 6 | 5 | 9
  Reticulocytes,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  Reticulocytes,DAY 1, PRE-DOSE,High | 0 | 0 | 0 | 1 | 0
  Reticulocytes,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  Reticulocytes,DAY 1, PRE-DOSE,Normal | 6 | 5 | 5 | 5 | 6
  Reticulocytes,DAY 1, PRE-DOSE,Missing: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  Reticulocytes,DAY 1, PRE-DOSE,Missing | 0 | 0 | 1 | 0 | 0
  Total Neutrophils,DAY 1, PRE-DOSE,High: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Neutrophils,DAY 1, PRE-DOSE,High | 0 | 1 | 1 | 1 | 0
  Total Neutrophils,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Neutrophils,DAY 1, PRE-DOSE,Normal | 5 | 5 | 6 | 4 | 6
  Total Neutrophils,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  Total Neutrophils,DAY 1 ,PRE-DOSE,Low | 1 | 0 | 0 | 1 | 0
  Total Neutrophils,DAY 1, 24 H,High: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Total Neutrophils,DAY 1, 24 H,High | 2 | 2 | 1 | 1 | 3
  Total Neutrophils,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 9 | 9 | 9 | 10
  Total Neutrophils,DAY 1, 24 H,Normal | 7 | 7 | 8 | 8 | 7
  WBC,DAY 1, PRE-DOSE,Normal: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  WBC,DAY 1, PRE-DOSE,Normal | 3 | 3 | 4 | 3 | 3
  WBC,DAY 1 ,PRE-DOSE,Low: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
  WBC,DAY 1 ,PRE-DOSE,Low | 3 | 3 | 3 | 3 | 3
  WBC,DAY 1, 24 H,Normal: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  WBC,DAY 1, 24 H,Normal | 8 | 7 | 8 | 9 | 7
  WBC,DAY 1, 24 H,Low: number analyzed (Participants) | 9 | 10 | 9 | 9 | 10
  WBC,DAY 1, 24 H,Low | 1 | 3 | 1 | 0 | 3

8. Primary Outcome: Summary of Urine Osmolality
Description: Urine sample was collected at screening, Day -2 (18:00h) and Day 1 (7:45h) for determination of urine osmolality which was measured in Millimole per kilogram (mmol/kg).
Time Frame: Day 1 (pre dose) of each treatment period
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/kg
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mmol/kg
  DAY -2: number analyzed (Participants) | 9 | 10 | 8 | 8 | 10
  DAY -2 | 631.8 (226.85) | 651.6 (229.44) | 647.1 (314.81) | 618.3 (314.15) | 702.2 (167.39)
  DAY 1,PRE-DOSE: number analyzed (Participants) | 6 | 5 | 6 | 4 | 6
  DAY 1,PRE-DOSE | 330.5 (88.89) | 364.4 (100.89) | 425.0 (257.05) | 304.3 (73.13) | 441.8 (87.61)

9. Primary Outcome: Mean Creatinine Clearance
Description: Creatinine clearance was calculated and reported in Milliliters per minute (mL/min) on Day 1 of each period for each collection interval 0-4, 4-8, 8-12, 12-16 and 16-24 hour, as well as the combined intervals of 0-12 and 0-24 hour. For urine measurements, participants were instructed to void within 30 minutes before administration of study medication.
Time Frame: Up to 24 hours post dose of each treatment period.
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mL/min
  0-4 H | 116.9 (43.28) | 134.5 (38.76) | 130.2 (44.13) | 142.2 (66.83) | 134.3 (61.43)
  4-8 H: number analyzed (Participants) | 10 | 10 | 10 | 10 | 9
  4-8 H | 111.5 (42.94) | 129.6 (54.27) | 122.7 (52.45) | 102.3 (31.01) | 134.0 (34.48)
  8-12 H: number analyzed (Participants) | 10 | 10 | 10 | 10 | 9
  8-12 H | 131.3 (63.82) | 123.3 (52.40) | 105.6 (37.92) | 140.6 (54.35) | 120.4 (43.29)
  12-16 H | 120.8 (49.47) | 117.9 (66.22) | 125.3 (78.45) | 89.5 (50.43) | 117.8 (61.66)
  16-24 H | 100.5 (40.47) | 119.5 (62.30) | 120.8 (33.73) | 126.4 (64.91) | 120.0 (33.91)
  0-12 H: number analyzed (Participants) | 10 | 10 | 10 | 10 | 9
  0-12 H | 119.9 (34.08) | 129.1 (28.34) | 119.5 (28.74) | 128.4 (37.85) | 132.7 (24.28)
  0-24 H: number analyzed (Participants) | 10 | 10 | 10 | 10 | 9
  0-24 H | 113.6 (30.30) | 124.0 (35.48) | 120.9 (30.05) | 121.3 (38.01) | 128.2 (26.45)

10. Primary Outcome: Summary of Fluid Balance
Description: On Day 1, fluid intake, urine volume and number of micturations were recorded over the intervals for each of the following dosing periods: 0-4h, 4-8h, 8-12h, 12-16h and 16-24h. From these measures, fluid balance was calculated over the 24-hour period. Fluid Balance=total fluid intake minus total urine volume. The 0-24h amounts of total Fluid Intake, total urine output, and fluid balance were calculated by adding the amounts collected during these time intervals.
Time Frame: Up to 24 hours post dose of each treatment period.
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Milliliters (mL)
  Total Fluid Intake,0-4h | 1240.0 (372.32) | 1274.4 (407.31) | 1221.0 (278.07) | 1009.5 (155.64) | 1201.0 (355.73)
  Total Fluid Intake,0-24h | 4196.3 (1399.83) | 4210.0 (1034.02) | 3934.7 (762.13) | 4164.4 (853.18) | 3998.2 (1110.77)
  Total urine output,0-4h | 1031.0 (277.04) | 1107.0 (294.54) | 1670.5 (451.39) | 1546.5 (593.86) | 1212.0 (424.94)
  Total urine output,0-24h | 4669.0 (757.00) | 4421.0 (741.14) | 5168.0 (1212.52) | 5004.0 (884.00) | 4941.0 (962.68)
  Fluid Balance,0-4h | 209.0 (352.43) | 167.4 (468.47) | -449.5 (533.77) | -537.0 (607.98) | -11.0 (541.71)
  Fluid Balance,0-24h | -472.7 (1076.26) | -211.0 (984.94) | -1233.3 (841.19) | -839.6 (772.69) | -942.8 (513.29)

11. Primary Outcome: Mean of Derived Plasma Glucose Parameters
Description: The plasma measurements at specified time points on Day 1 were collected. Derived plasma glucose parameters were presented.
Time Frame: Up to 24 hours post dose of each treatment period.
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mmol/L
  Pre-Dose | 5.75639 (1.285496) | 6.65953 (1.165222) | 6.18659 (1.696588) | 5.72419 (0.850452) | 5.86796 (0.881584)
  2 h | 18.26279 (2.222558) | 13.70542 (4.831705) | 16.11455 (3.711572) | 14.76566 (2.542980) | 15.00435 (3.158931)
  4 h | 15.31521 (3.646185) | 9.47778 (4.288005) | 11.52943 (3.154919) | 10.68068 (3.161241) | 11.04094 (3.184558)
  6 h | 19.53952 (4.101401) | 9.91464 (3.978186) | 16.02019 (4.685123) | 14.97660 (5.647356) | 15.50949 (4.792842)
  8 h | 18.01300 (5.158167) | 8.87790 (2.958162) | 14.21611 (5.359803) | 13.69432 (6.375146) | 14.47146 (5.477677)
  12 h | 14.67129 (6.061024) | 11.34791 (3.897886) | 12.95048 (4.566692) | 11.31849 (3.376891) | 11.87914 (4.053962)

12. Secondary Outcome: Incremental Adjusted Weighted Means of Plasma Glucose AUC(0-4) and AUC(0-10) on Day 1
Description: AUC(0-10) was the plasma glucose weighted mean AUC for 0 to 10 h post-dosing and AUC(0-4) was the plasma glucose weighted mean AUC for 0 to 4 h post-dosing. Incremental Adjusted Weighted Means were presented.
Time Frame: Up to 24 hours post dose of each treatment period.
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mmol/L
  AUC(0-4) | 8.739 (2.4304) | 4.480 (2.9942) | 6.632 (2.0126) | 6.044 (1.9444) | 6.099 (2.3135)
  AUC(0-10) | 10.535 (3.8388) | 3.127 (2.2467) | 7.112 (3.3103) | 6.653 (3.2809) | 7.054 (3.5440)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 50mg; Difference from placebo to GSK189075 50mg AUC(0-4) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0008, ANCOVA; Median Difference (Final Values) = -2.728, 95% CI 2-sided [-4.219 to -1.236]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 150mg; Difference from placebo toGSK189075 150mg AUC(0-4) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0021, ANCOVA; Mean Difference (Final Values) = -2.325, 95% CI 2-sided [-3.735 to -0.916]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500mg; Difference from placebo to GSK189075 500mg AUC(0-4) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0021, ANCOVA; Mean Difference (Final Values) = -2.402, 95% CI 2-sided [-3.862 to -0.942]
Statistical Analysis 4: Comparison: Placebo+ Prandial Insulin vs GSK189075 50mg; Difference from Placebo+ Prandial insulin to GSK189075 50mg AUC(0-4) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0382, ANCOVA; Mean Difference (Final Values) = 1.556, 95% CI 2-sided [0.090 to 3.021]
Statistical Analysis 5: Comparison: Placebo+ Prandial Insulin vs GSK189075 150mg; Difference from Placebo+ Prandial insulin to GSK189075 150mg AUC(0-4) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0132, ANCOVA; Mean Difference (Final Values) = 1.958, 95% CI 2-sided [0.439 to 3.477]
Statistical Analysis 6: Comparison: Placebo+ Prandial Insulin vs GSK189075 500mg; Difference from Placebo+ Prandial insulin to GSK189075 500mg AUC(0-4) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0161, ANCOVA; Mean Difference (Final Values) = 1.881, 95% CI 2-sided [0.373 to 3.389]
Statistical Analysis 7: Comparison: Placebo vs GSK189075 50mg; Difference from placebo to GSK189075 50mg AUC(0-10) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Net) = -3.592, 95% CI 2-sided [-5.162 to -2.022]
Statistical Analysis 8: Comparison: Placebo vs GSK189075 150mg; Difference from placebo to GSK189075 150mg AUC(0-10) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0000, ANCOVA; Mean Difference (Final Values) = -3.820, 95% CI 2-sided [-5.304 to -2.337]
Statistical Analysis 9: Comparison: Placebo vs GSK189075 500mg; Difference from placebo to GSK189075 500mg AUC(0-10) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -2.887, 95% CI 2-sided [-4.424 to -1.350]
Statistical Analysis 10: Comparison: Placebo+ Prandial Insulin vs GSK189075 50mg; Difference from Placebo+ Prandial insulin to GSK189075 50mg AUC(0-10) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 2.953, 95% CI 2-sided [1.411 to 4.496]
Statistical Analysis 11: Comparison: Placebo+ Prandial Insulin vs GSK189075 150mg; Difference from Placebo+ Prandial insulin to GSK189075 150mg AUC(0-10) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0015, ANCOVA; Mean Difference (Final Values) = 2.725, 95% CI 2-sided [1.126 to 4.324]
Statistical Analysis 12: Comparison: Placebo+ Prandial Insulin vs GSK189075 500mg; Difference from Placebo+ Prandial insulin to GSK189075 500mg AUC(0-10) Incremental Adjusted Weighted Mean; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = 3.659, 95% CI 2-sided [2.071 to 5.246]

13. Secondary Outcome: Urinary Glucose Excretion (UGE) for Timed Subintervals up to 24 Hours Post Dose (0-24 H)
Description: UGE was assessed for timed subintervals up to 24h post-dose. Urine samples were collected at intervals: 0-4h, 4-8h, 8-12h, 12-16h and 16-24h on study days. The 0-24h amounts excreted in urine were calculated by adding the amounts collected during these time intervals.
Time Frame: Up to 24 hours post dose of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mmol | 324.849 (252.6604) | 135.119 (191.6857) | 579.060 (227.9230) | 601.879 (206.4860) | 770.249 (245.1817)

14. Secondary Outcome: Percent of Filtered Glucose in the Urine.
Description: Filtered glucose in the urine was assessed at indicated time points and was presented as Percentage. The 0-12h and 0-24h amounts Percent of filtered glucose in the urine were calculated by adding the amounts collected during these time intervals.
Time Frame: Up to 24 hours post dose of each treatment period.
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Percentage
  0-4 H | 10.8661 (6.21239) | 6.5576 (5.24295) | 40.4788 (7.00049) | 41.5290 (14.95891) | 41.3449 (12.49532)
  0-12 H | 16.7543 (9.04186) | 7.0663 (8.62344) | 42.3900 (5.75325) | 47.5648 (10.41524) | 47.8442 (12.01952)
  0-24 H | 11.1012 (5.76206) | 5.6518 (5.12934) | 25.4355 (4.74207) | 29.9386 (5.99518) | 34.5245 (10.00663)

15. Secondary Outcome: Mean Total Urine Volume 0-24 H
Description: Urine volume was recorded over intervals : 0-4h, 4-8h, 8-12h, 12-16h and 16- 24h on Day 1 for each dosing period. Mean total Urine volume over 24 hours was presented.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mL | 4628.5 (746.74) | 4623.0 (828.93) | 5267.5 (1077.76) | 4962.0 (885.86) | 5274.4 (899.07)

16. Secondary Outcome: Mean Creatinine Clearance 0-24 H
Description: Urine samples for calculating creatinine clearance were obtained over the intervals: 0-4h, 4-8h, 8-12h, 12-16h and 16-24h. Mean creatinine clearance over 0-24 H was presented.
Time Frame: Day 1 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mL/min | 113.6 (30.30) | 124.0 (35.48) | 120.9 (30.05) | 121.3 (38.01) | 128.2 (26.45)

17. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUC) From Time Zero (Time of Dosing) to the Last Time Point With Measurable Analyte Concentration, AUC(0-last), AUC From Time Zero to Infinite Time, AUC(0-inf) of GSK189075 Over Period
Description: AUC(0-last) was defined as area under the plasma concentration vs. time curve from time zero (time of dosing) to the last time point with measurable analyte concentration and AUC(0-inf) was defined as area under the plasma concentration vs. time curve from time zero to infinite time. Blood samples were collected on time points: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period.
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (hr*ng/mL)
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
hour*nanograms per milliliter (hr*ng/mL)
  AUC(0-inf) | 8.101 (24) | 25.922 (38) | 58.362 (60)
  AUC(0-last) | 3.966 (95) | 16.552 (57) | 47.390 (67)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK189075 Over Period
Description: Plasma samples for pharmacokinetic analysis were drawn at indicated time points of each treatment period. Cmax was defined as maximal measured plasma concentration over the time span specified. Values were reported as Geometric Means with respective Geometric Coefficient of Variation (% CV).
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
ng/mL | 5.266 (90) | 11.903 (92) | 39.029 (128)

19. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) and Terminal Half Life, (T1/2) of GSK189075 Over Period
Description: Tmax was defined as the time to the maximum or "peak" concentration of a drug observed after multiple administration. T1/2 was defined as the time to when half of the total amount of a particular substance is eliminated from the body. Blood samples obtained during indicated time points. T1/2 was calculated as t1/2 = ln2/λz, with λz (the terminal elimination rate-constant) estimated from log-linear regression analysis of the terminal phase of the plasma concentration-time profile.Tmax and t1/2 values for GSK189075 were presented.
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Safety Population. Only those participants available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
hour
  Tmax | 0.446 (68) | 0.521 (81) | 1.054 (145)
  t1/2: number analyzed (Participants) | 5 | 5 | 5
  t1/2 | 0.915 (20) | 1.019 (41) | 0.678 (29)

20. Secondary Outcome: AUC From Time Zero to 4 Hours Post Dose, AUC(0-4) for GSK189074 Over Period
Description: AUC(0-4) was defined as AUC from time zero to 4 hours post dose. Blood samples were collected on time points: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period.
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
hr*ng/mL | 243.281 (34) | 700.970 (38) | 2038.298 (34)

21. Secondary Outcome: Oral Clearance (CL/F) Over Period
Description: Oral clearance is a measure of the rate at which the drug is cleared from the body via metabolism. Blood samples were collected on time points: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
mL/min | 2849.947 (36) | 2732.322 (41) | 2903.590 (37)

22. Secondary Outcome: The Metabolite to Parent AUC Ratio, AUCmetabolite/AUCparent Ratio for GSK189074 Over Period
Description: Blood samples were collected on time points: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period to obtain the metabolite to parent AUC ratio for GSK189074
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
Ratio | 90.436 (70) | 67.801 (36) | 74.281 (52)

23. Secondary Outcome: The Metabolite to Parent AUC Ratio, AUCmetabolite/AUCparent Ratio for GSK279782 Over Period
Description: Blood samples were collected on time points: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period to obtain the metabolite to parent AUC ratio for GSK279782
Time Frame: Pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h of each treatment period
Population: Pharmacokinetic (PK) Parameter Population comprised of all participants for whom pharmacokinetic parameter estimates were derived during any treatment period
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
Number analyzed (Participants) | 10 | 10 | 10
Ratio | 0.427 (58) | 0.442 (60) | 0.433 (55)

ADVERSE EVENTS:
Time Frame: Approximately up to 6 months
Description: Safety population was used.
Arm/Group | Placebo | Placebo+ Prandial Insulin | GSK189075 50mg | GSK189075 150mg | GSK189075 500mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 4/10 | 5/10 | 6/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Placebo+ Prandial Insulin (N=10) | GSK189075 50mg (N=10) | GSK189075 150mg (N=10) | GSK189075 500mg (N=10)
Headache (Nervous system disorders) | 2 | 2 | 3 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.